CLINICAL TRIAL: NCT00525499
Title: A Phase 2, Multi-Center, Randomized, Double-Blind, Vehicle-Controlled Dose-Ranging Clinical Study to Evaluate the Safety and Efficacy of ASC-J9 Cream Applied Twice Daily for 12 Weeks for the Treatment of Facial Acne Vulgaris
Brief Title: A Phase 2 Study of ASC-J9 Cream in Acne Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AndroScience Corp (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASC-J9-201
Record Dates: First submitted 2007-08-31; First posted 2007-09-05 (Estimated); Results first posted 2011-04-18 (Estimated); Last update posted 2011-11-23 (Estimated); Status verified 2011-11

CONDITIONS: Acne Vulgaris
Keywords: acne
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Placebo Comparator): Vehicle control cream applied topically to the face twice daily for 12 weeks
  Interventions: Drug: placebo
- 2 (Experimental): 0.001% ASC-J9 cream applied topically to the face twice daily for 12 weeks
  Interventions: Drug: ASC-J9 cream
- 3 (Experimental): 0.005% ASC-J9 cream applied topically to the face twice daily for 12 weeks
  Interventions: Drug: ASC-J9 cream
- 4 (Experimental): 0.025% ASC-J9 cream applied topically to the face twice daily for 12 weeks
  Interventions: Drug: ASC-J9 cream

INTERVENTIONS:
Drug: ASC-J9 cream — Topical application to the face twice daily for 12 weeks.
  Arms: 2; 3; 4
Drug: placebo — vehicle control applied topically twice daily for 12 weeks
  Other Names: Androgen receptor degradation enhancer
  Arms: 1

SUMMARY:
The purpose of this study is to evaluate if topical ASC-J9 cream is effective in treating acne.

DETAILED DESCRIPTION:
Subjects with acne were randomized to one of four treatment groups for twice daily topical dosing to the face for 12 weeks. Assessments of acne status were performed at Baseline, Weeks 2, 4, 8 and 12 and then 4 weeks after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* At least 12 years of age.
* Facial acne, with:

  20 -100 inflammatory facial lesions 20 -100 noninflammatory facial lesions No more than 2 nodules/cysts on the face

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Skin diseases other than acne vulgaris
* Use of oral retinoids within 6 months of Baseline Visit
* Unwilling to discontinue all other treatments for facial acne
* Unwilling to avoid excessive swimming/sun exposure and use of cosmetics

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2007-08; Primary Completion 2008-04 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles CY Shih, PhD, Study Chair — AndroScience Corp
Locations (10):
- United States (10):
  - East Bay Dermatology Medical Group, Fremont, California
  - Therapeutics Clinical Research, San Diego, California
  - Northwest Clinical Trial, Boise, Idaho
  - TKL Research, Inc, Paramus, New Jersey
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - Dermatology Associates, Knoxville, Tennessee
  - DermResearch, Inc, Austin, Texas
  - J&S Studies, Inc, Bryan, Texas
  - Dermatology Research Center, Inc, Salt Lake City, Utah
  - Education and Research Foundation, Lynchburg, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Vehicle Control: Vehicle control cream applied topically to the face twice daily for 12 weeks
- 0.001% ASC-J9 Cream: 0.001% ASC-J9 cream applied topically to the face twice daily for 12 weeks
- 0.005% ASC-J9 Cream: 0.005% ASC-J9 cream applied topically to the face twice daily for 12 weeks
- 0.025% ASC-J9 Cream: 0.025% ASC-J9 cream applied topically to the face twice daily for 12 weeks
Period: Overall Study
Arm/Group | Vehicle Control | 0.001% ASC-J9 Cream | 0.005% ASC-J9 Cream | 0.025% ASC-J9 Cream
Started | 47 | 46 | 47 | 46
Completed | 40 | 39 | 40 | 39
Not Completed | 7 | 7 | 7 | 7
Not completed — Lost to Follow-up | 2 | 4 | 1 | 4
Not completed — Adverse Event | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 5 | 1 | 5 | 2
Not completed — Protocol Violation | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vehicle Control | 0.001% ASC-J9 Cream | 0.005% ASC-J9 Cream | 0.025% ASC-J9 Cream | Total
Number analyzed (Participants) | 47 | 46 | 47 | 46 | 186
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 33 | 33 | 32 | 31 | 129
  Between 18 and 65 years | 14 | 13 | 15 | 15 | 57
  >=65 years | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 17.7 (4.9) | 18.0 (4.9) | 17.7 (5.8) | 18.3 (5.3) | 17.9 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 27 | 19 | 16 | 76
  Male | 33 | 19 | 28 | 30 | 110
Region of Enrollment [Number; unit: participants]
  United States | 47 | 46 | 47 | 46 | 186

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Inflammatory Acne Lesion Counts From Baseline to Week 12
Description: Percent change in inflammatory lesion counts from Baseline to Week 12. It is calculated by taking the Week 12 count minus the Baseline count and then dividing by the Baseline count. Thus, a negative percent change will reflect a reduction in lesion counts.
Time Frame: Baseline to Week 12
Population: ITT population: All randomized subjects
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Vehicle Control | 0.001% ASC-J9 Cream | 0.005% ASC-J9 Cream | 0.025% ASC-J9 Cream
Number analyzed (Participants) | 47 | 46 | 47 | 46
Percent change | -37.4 (41.0) | -34.7 (32.4) | -30.7 (47.6) | -44.8 (35.6)

2. Secondary Outcome: Number of Participants With Improvement in Investigator Global Assessment by at Least One Grade From Baseline to Week 12
Description: The Investigator Global Assessment used a static categorical scale, with zero corresponding to no acne and higher scores reflecting more severe acne:
  0 No acne lesions.
  1. Rare non-inflammatory lesions.
  2. Some non-inflammatory lesions, no more than a few inflammatory lesions. No nodulo-cystic lesions.
  3. Many non-inflammatory lesions, some inflammatory lesions, no more than one nodulo-cystic lesion.
  4. Many noninflammatory and inflammatory lesions but no more than a few nodulo-cystic lesions.
  5. Highly inflammatory lesions, multiple nodulo-cystic lesions.
Time Frame: Baseline to Week 12
Population: ITT population: All randomized subjects
Measure: Number; unit: Participants
Arm/Group | Vehicle Control | 0.001% ASC-J9 Cream | 0.005% ASC-J9 Cream | 0.025% ASC-J9 Cream
Number analyzed (Participants) | 47 | 46 | 47 | 46
Participants | 23 | 20 | 23 | 28

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Vehicle Control | 0.001% ASC-J9 Cream | 0.005% ASC-J9 Cream | 0.025% ASC-J9 Cream
Serious Adverse Events (participants affected / at risk) | 1/47 | 0/46 | 0/47 | 0/46
Other Adverse Events (participants affected / at risk) | 5/47 | 11/46 | 8/47 | 14/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle Control (N=47) | 0.001% ASC-J9 Cream (N=46) | 0.005% ASC-J9 Cream (N=47) | 0.025% ASC-J9 Cream (N=46)
Viral meningitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle Control (N=47) | 0.001% ASC-J9 Cream (N=46) | 0.005% ASC-J9 Cream (N=47) | 0.025% ASC-J9 Cream (N=46)
nasopharyngitis (Infections and infestations) | 4 (4) | 4 (4) | 6 (6) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 6 (6) | 1 (1) | 6 (6)
Streptococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Institution and Investigator agree not to publish the results of this study without the prior written consent of Sponsor.